CLINICAL TRIAL: NCT01629394
Title: Comparative Study of Sugammadex Versus Neostigmine for Reversal of Neuromuscular Blockade in Morbidly Obese Patients Undergoing Weight Loss Surgery.Use of Acceleromyography Monitoring in Adductor Pollicis and Corrugator Supercilii.
Brief Title: Comparative Study of Sugammadex Versus Neostigmine for Reversal of Neuromuscular Blockade in Morbidly Obese Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Prokopios Georgiou, Prokopios Georgiou M.D., University of Patras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 952/21-3-12
Record Dates: First submitted 2012-04-01; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Morbid Obesity; Neuromuscular Blockade
MeSH Terms: conditions — Obesity, Morbid | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group A: Sugammadex CBW-open (Active Comparator): Group A patients will undergo open surgery and will receive sugammadex 2mg/kg corrected body weight [corrected body weight = ideal body weight + 40%( real body weight - ideal body weight)] when T2 arises in adductor pollicis.
  Interventions: Drug: Sugammadex
- Group B: Sugammadex IBW-open (Active Comparator): Group B patients will undergo open surgery and will receive sugammadex 2mg/kg ( ideal body weight ) when T2 arises in adductor pollicis.
  Interventions: Drug: Sugammadex
- Group C: Neostigmine CBW-open (Active Comparator): Group C patients will undergo open surgery and will receive neostigmine 50μg/kg corrected body weight [corrected body weight = ideal body weight + 40%(real body weight - ideal body weight)]when T2 arises in adductor pollicis.
  Interventions: Drug: Neostigmine
- Group D: Neostigmine-IBW (Active Comparator): Group D patients will undergo open surgery and will receive neostigmine 50μg/kg ( ideal body weight ) when T2 arises in adductor pollicis.
  Interventions: Drug: Neostigmine
- Group E: Sugammadex CBW-Lap (Active Comparator): Group E patients will undergo laparoscopic surgery and will receive sugammadex 2mg/kg corrected body weight [corrected body weight = ideal body weight + 40%( real body weight - ideal body weight)] when T2 arises in adductor pollicis.
  Interventions: Drug: Sugammadex
- Group F: Sugammadex IBW-Lap (Active Comparator): Group F patients will undergo laparoscopic surgery and will receive sugammadex 2mg/kg ( ideal body weight ) when T2 arises in adductor pollicis.
  Interventions: Drug: Sugammadex
- Group G: Neostigmine CBW-Lap (Active Comparator): Group C patients will undergo laparoscopic surgery and will receive neostigmine 50μg/kg corrected body weight [corrected body weight = ideal body weight + 40%(real body weight - ideal body weight)]when T2 arises in adductor pollicis.
  Interventions: Drug: Neostigmine
- Group H: Neostigmine IBW-Lap (Active Comparator): Group D patients will undergo open surgery and will receive neostigmine 50μg/kg ( ideal body weight ) when T2 arises in adductor pollicis.
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Single dose of 2 mg/kg corrected body weight [corrected body weight = ideal body weight + 40%(real body weight - ideal body weight)]
  Other Names: Bridion(R)
  Arms: Group A: Sugammadex CBW-open
Drug: Sugammadex — Single dose of sugammadex 2 mg/kg ( ideal body weight )
  Other Names: Bridion(R)
  Arms: Group B: Sugammadex IBW-open
Drug: Neostigmine — Single dose of neostigmine 50 μg/kg corrected body weight [corrected body weight = ideal body weight + 40%(real body weight - ideal body weight)]
  Arms: Group C: Neostigmine CBW-open
Drug: Neostigmine — Single dose of neostigmine 50 μg/kg ( ideal body weight )
  Arms: Group D: Neostigmine-IBW
Drug: Sugammadex — Single dose of 2 mg/kg corrected body weight [corrected body weight = ideal body weight + 40%( real body weight - ideal body weight)]
  Other Names: Bridion(R)
  Arms: Group E: Sugammadex CBW-Lap
Drug: Sugammadex — Single dose of sugammadex 2 mg/kg ( ideal body weight )
  Other Names: Bridion(R)
  Arms: Group F: Sugammadex IBW-Lap
Drug: Neostigmine — Single dose of neostigmine 50 μg/kg corrected body weight [corrected body weight = ideal body weight + 40%(real body weight - ideal body weight)]
  Arms: Group G: Neostigmine CBW-Lap
Drug: Neostigmine — Single dose of neostigmine 50μg/kg ( ideal body weight )
  Arms: Group H: Neostigmine IBW-Lap

SUMMARY:
Postoperative residual curarization in the post anaesthesia unit has been associated to complications involving respiratory function and impaired laryngeal and pharyngeal muscles' function. Speed of reversal of neuromuscular blockade after administration of sugammadex versus neostigmine has been studied, but up to date no data are available concerning continuous acceleromyography monitoring of adductor pollicis and corrugator supercilii in morbidly obese patients undergoing weight loss surgery. The investigators' aim in this prospective, double-blinded study was to compare train of four ( TOF ) values, the presence or absence of clinical criteria of postoperative residual curarization , the dose requirements and the side effects of sugammadex and neostigmine for the reversal of rocuronium induced neuromuscular blockade in patients undergoing laparoscopic or open surgery for morbid obesity.

DETAILED DESCRIPTION:
Morbidly obese patients [ body mass index (BMI) > 40 kg/m2 ] planned to undergo open or laparoscopic surgery for weight loss will be managed with standardized general anesthesia (intravenous Propofol combined with remifentanil and muscle relaxation induced by rocuronium).

By the end of the surgery, Group A and group E patients will receive sugammadex 2 mg/kg corrected body weight [corrected body weight(CBW)=ideal body weight(IBW) + 40%(real body weight(RBW)-ideal body weight)] when T2 arises in adductor pollicis. Group C and group G will receive neostigmine 50μg/kg corrected body weight when T2 arises in adductor pollicis. Group B and group F patients will receive sugammadex 2 mg/kg ideal body weight when T2 arises in adductor pollicis. Group D and group H patients will receive 50μg/kg neostigmine ideal body weight.

Investigators will proceed in continuous acceleromyography monitoring of adductor pollicis and corrugator supercilii during induction of anaesthesia, surgery, recovery and in the post anaesthesia care unit, recording TOF values. Total consumption of neuromuscular blocking agent, doses of reversal agents and clinical criteria of post operation residual curarization will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >40kg
* Age < 60
* Patients written consent to participate in the study

Exclusion Criteria:

* Cardiovascular disease (NYHA>2)
* Patients refusal to participate in the study
* Contraindication to epidural catheter placement (e.g anticoagulation, anti- platelets medication)
* coexisting neuromuscular disease
* history of allergic reaction to neuromuscular blocking agents
* history of difficult intubation
* creatinine levels > 159lmol/l

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Speed of reversal of neuromuscular blockade after administration of different sugammadex/neostigmine doses to TOF values = 0.9 in adductor pollicis and corrugator supercilii | TOF values for 2.5 h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Prokopios S. Georgiou, M.D., Principal Investigator — University Hospital of Patras; Kriton S. Filos, Professor, Study Chair — University of Patras, Dept. of Anaesthesiology and Critical Care Medicine; Athena Siampalioti, M.D., Study Director — University Hospital of Patras
Locations (1):
- University of Patras, Department of Anesthesiology and Critical Care Medicine, Pátrai, Achaia, Greece